CLINICAL TRIAL: NCT03833726
Title: Light Emitting Diode for the Treatment of Genitourinary Syndrome of Menopause Associated With Hormonal Therapy for Treating Breast Cancer: Randomized Controlled Clinical Trial
Brief Title: Light Emitting Diode for theTreatment of Genitourinary Syndrome of Menopause Associated With Breast Cancer Treatment
Acronym: LEDCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAP CA
Record Dates: First submitted 2018-12-16; First posted 2019-02-07 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Atrophy;Vaginal; Breast Cancer
Keywords: Vaginal Atrophy; Breast Cancer; Hormonal Therapy; Photodynamic Therapy; Light Emitting Diode
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will be conducted women diagnosed with Genitourinary Syndrome of Menopause treated with kinesiotherapy, divided in two groups: LED treatment or LED Sham.
Who Masked: Participant, Care Provider
Masking Description: The participant will be randomly divided between LED group or LED Sham procedure that will consist of turned off device and heated gel and both patients and physiotherapists of kinesiotherapy phase wont be aware with group the participant is allocated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LED group (Experimental): Participants who will submitted to active procedure with LED. Both groups will be submitted to kinesiotherapy.
  Interventions: Procedure: Experimental: LED group
- Control group (Sham Comparator): Participants who will submitted to sham procedure with heated gel. Both groups will be submitted to kinesiotherapy.
  Interventions: Procedure: Sham Comparator: Control

INTERVENTIONS:
Procedure: Experimental: LED group — 5 Sessions of 8 minute 405 nm Blue Light Emitting Diode, LED, with a power of 1.66 W / m2, 7 days apart.
  Arms: LED group
Procedure: Sham Comparator: Control — 5 Sessions of 8 minute with device off and heated gel, 7 days apart.
  Arms: Control group

SUMMARY:
Breast Cancer treatment may cause several side effects, some long lasting. Adjuvant hormone therapy helps avoiding recurrence triggers vulvovaginal atrophy syndrome. This study evaluate a photodynamic treatment with light emitting diode to improve vaginal dryness and irritation, pruritus, pain or discomfort in intercourse.

DETAILED DESCRIPTION:
The Genitourinary Menopause Syndrome (MMS) affects up to 70% of in treatment breast cancer patients. Symptoms are due to a decrease in hormone levels or block to circulating hormones and induce functional changes in the vagina cutting in quality of life and impacting sexual function.

This is a randomized, double blind trial in a sample of 74 individuals that will be performed at an specialized Pelvic Floor Care Center (CAAP) in Brazil. Will be included women age between 18 and 65 years, in adjuvant hormone therapy, with clinical signs and symptoms of vulvovaginal atrophy syndrome and cytologic evidence of atrophy, (pH <5.0 and vaginal cytology with predominance of superficial cells).

Will be excluded from the study the patients in hormonal replacement for less than 6 months, diagnosis of vaginal infection, pregnant women, difficulty understanding the proposed instruments and patients with chronic neurological degenerative diseases.

Three 405 nm light emitting diode (LED) sessions will be performed, with a seven days interval between them compared with sham procedure, and both groups will perform five sessions of kinesiotherapy sessions.

Maturation vaginal index will be checked before and after all treatment and self- administered questionnaires will be performed before each session with Female Sexual Function Index (FSFI) - Female Version (QS-F), Female Genital Self-Image Scale - 7 (FGSIS-7), International Consultation on Incontinence Questionnaire - Short Form, (ICIQ-SF), Functional Assessment Of Cancer Therapy - Breast Cancer (FACT-B).

At the end of treatment, the visual analog scale and Likert scale will be used to measure the individual's satisfaction

ELIGIBILITY:
Inclusion Criteria:

* 18-65 anos
* Pathological proven Breast Cancer diagnosis
* Stage 0-III by American Joint Committee on Cancer (AJCC) and International Union Against Cancer (UICC) of Classification of Malignant Tumours, TNM (Acronym for Tumor-Node-Metastasis) 8ª edition
* Genitourinary Syndrome of Menopause confirmed through patient-reported symptoms and gynecological examination (of external structures, introitus, and vaginal mucosa)
* Vaginal pH >5,0

Exclusion Criteria:

* Hormone replacement less than 6 months
* Diagnosis of vaginal infection
* Difficulty in understanding the proposed instruments
* Patients with chronic neurological degenerative diseases that preclude to be on position
* Metastatic disease
* Any vaginal photodynamic treatment less than 3 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Vaginal maturation index | Change from baseline at 3 months
  Cytological vaginal will be collected at 1/3 lower lateral vaginal wall and quantified superficial, intermediate and basal cells to calculate vaginal maturation index
Female Sexual Function Index (FSFI) - Female Version (QS-F) | Change from baseline at 3 months
  Measure of quality of sex life. Full Scale Score Range 2-36

SECONDARY OUTCOMES:
Vaginal pH | Change from baseline at 3 months
  pH indicator tape
Quality of life by FACT B | Change from baseline at 3 months
  Functional Assessment of Chronic Therapy- Breast (FACT B) Questionary validated to Portuguese to measure quality of life in breast cancer patients (Total score and Subscale). Graduated 0-128 (lower values means worse quality of life). Physical Wellbeing (PWB) 0-28; Social/Family Wellbeing (SWB) 0-28; Emotional Wellbeing (EWB) 0-24; Funtional Wellbeing (FWB) 0-28; Breast Cancer Subscale (BCS) 0-40. Total Score do not include Arm Subscale (ARM) 0-20
Urinary symptoms | Change from baseline at 3 months
  International Consultation on Incontinence Questionnaire - Short Form (ICIQ Questionary Short Form)-Scoring scale: 0-21 (lower values means better quality of life)
Visual analog scale | Change from baseline at 3 months
  Stratification between 0 and 10 (few symptoms to severe symptoms)
Female Genital Self-Image Scale - 7 (FGSIS-7) | Change from baseline at 3 months
  Measure of quality of sex life. Scores between 7-28 (higher scores indicate better self-image)
Likert scale | Change from finished treatment and 3 months after
  Satisfaction with the treatment measured between 1 and 5 ( not at all happy with the treatment -very happy with the treatment)
Sexual Quotients Female Version (QS-F) | Change from baseline at 3 months
  Female sex life domain. Scores between 0-100 (higher scores indicate better sex life) Scores between 82-100 score: excellent, 62-80 score: regular, 42-60 score: unfavorable, 22-40 score: regular, 0-20 score: bad
SF-36 | Change from baseline at 3 months
  Short Form health survey 36 questionnaire, (0-100) - lower values means worse quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Patríca V Lordelo, PhD, Study Chair — Centro de Atenção Pélvica- CAAP
Locations (1):
- Centro de Atenção ao Assoalho Pelvico, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Background] Lester J, Pahouja G, Andersen B, Lustberg M. Atrophic vaginitis in breast cancer survivors: a difficult survivorship issue. J Pers Med. 2015 Mar 25;5(2):50-66. doi: 10.3390/jpm5020050. PMID 25815692
- [Background] Kyvernitakis I, Ziller V, Hars O, Bauer M, Kalder M, Hadji P. Prevalence of menopausal symptoms and their influence on adherence in women with breast cancer. Climacteric. 2014 Jun;17(3):252-9. doi: 10.3109/13697137.2013.819327. Epub 2013 Aug 25. PMID 23805799
- [Background] Portman DJ, Gass ML; Vulvovaginal Atrophy Terminology Consensus Conference Panel. Genitourinary syndrome of menopause: new terminology for vulvovaginal atrophy from the International Society for the Study of Women's Sexual Health and the North American Menopause Society. Maturitas. 2014 Nov;79(3):349-54. doi: 10.1016/j.maturitas.2014.07.013. Epub 2014 Aug 19. PMID 25179577
- [Background] Nilsson K, Risberg B, Heimer G. The vaginal epithelium in the postmenopause--cytology, histology and pH as methods of assessment. Maturitas. 1995 Jan;21(1):51-6. doi: 10.1016/0378-5122(94)00863-3. PMID 7731384
- [Background] Moreno AC, Sikka SK, Thacker HL. Genitourinary syndrome of menopause in breast cancer survivors:Treatments are available. Cleve Clin J Med. 2018 Oct;85(10):760-766. doi: 10.3949/ccjm.85a.17108. PMID 30289755
- [Background] Arunkalaivanan A, Kaur H, Onuma O. Laser therapy as a treatment modality for genitourinary syndrome of menopause: a critical appraisal of evidence. Int Urogynecol J. 2017 May;28(5):681-685. doi: 10.1007/s00192-017-3282-y. Epub 2017 Feb 2. PMID 28154914
- [Background] Yaralizadeh M, Abedi P, Najar S, Namjoyan F, Saki A. Effect of Foeniculum vulgare (fennel) vaginal cream on vaginal atrophy in postmenopausal women: A double-blind randomized placebo-controlled trial. Maturitas. 2016 Feb;84:75-80. doi: 10.1016/j.maturitas.2015.11.005. Epub 2015 Nov 12. PMID 26617271
- See also: NCI Toxicity Scale — http://evs.nci.nih.gov/ftp1/CTCAE